CLINICAL TRIAL: NCT03757832
Title: Feasibility Study to Estimate Fat Concentration of Liver in Adults Through RF Imaging
Brief Title: Fatty Liver Imaging Project
Acronym: FLIP
Status: Completed | Type: Observational
Sponsor: Aaron Fenster (Other)
Responsible Party: Sponsor-Investigator, Aaron Fenster, Scientist, Western University, Canada
Organization: Western University, Canada (Other)
Other Study IDs: 111117
Record Dates: First submitted 2018-11-27; First posted 2018-11-29 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Determine the Number of Anatomical Sites at Which Successful Thermoacoustic Fat Measurements Can be Made From Five Acquisitions Using the FLIP ITA Device; Determine the Correlation of Fat Measures Obtained by the FLIP Device and Those Obtained From Quantitative MRI; Provide Insight Into the Sensitivity of Thermoacoustic Liver Fat Assessment With the Aim of Detecting Fat Content in Liver at 15% or Less, by Volume

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Liver Imaging — The device will acquire thermoacoustic data while the ultrasound probe acquires ultrasound images, and an MR of the liver is acquired as a comparative modality.

SUMMARY:
This study is being done to test the FLIP device, a novel device developed and manufactured by Endra Life Sciences, located in Ann Arbor, Michigan. The purpose of the device is to measure the fat content of liver tissue to assist in the diagnosis of fatty liver disease. This feasibility study will involve 25 healthy volunteers having their liver imaged by traditional ultrasound and MRI methods as well as using the FLIP device. The data obtained by the FLIP will be compared with the data obtained by ultrasound and MRI in order to determine the effectiveness of the device. This is a preliminary study to see if the investigational device could eventually be used to image the liver alongside traditional ultrasound for discerning fat concentration.

DETAILED DESCRIPTION:
It has been demonstrated that thermoacoustic imaging can be used to identify water and fat concentrations [Bauer, 2012]. In addition, the group led by Dr. Kruger have demonstrated that conventional computed tomography shows similar features to thermoacoustic imaging in small animal studies [Kruger, 2003]. These concepts have led Endra Life Sciences to develop the FLIP device with the purpose of imaging fat concentration in liver tissue with indications for fatty liver disease. Non-alcoholic fatty liver disease (NAFLD) was first reported in 1980 by pathologists at the Mayo clinic in obese, or overweight, patients with no history of alcohol abuse. This represented the first time that fatty livers were observed with no history of alcohol abuse. Since that first report of NAFLD, increased rates of obesity and general increased caloric intake has dramatically increased rates of fatty liver disease. Estimates of NAFLD range from 25 - 40% of the adult population globally. NAFLD is a multi-system disease. Fatty liver disease is highly correlated with obesity and alcohol abuse, and is an important biomarker of insulin resistance and metabolic disease. Endra's technology offers a non-invasive, cost effective point of care solution to monitoring liver fat content that will be enormously helpful in surveilling patients with metabolic disease, insulin resistance, and those at risk for later stage liver disease.

This study will provide additional information that will guide the further development of the FLIP device with the end goal of commercializing the product. Fibroscan is a device that is currently on the market that is also indicated for fatty liver disease. Fibroscan is a shear wave elastography device that measures the stiffness of liver tissue by mechanically deforming tissue (by utilizing a plunger that vibrates the surface of the skin) and measures the resulting shear wave speed within the liver by ultrasound. The shear wave speed is related to the mechanical stiffness of the tissue. Fibroscan aims to assess the progression of infiltration of collagen into normal liver tissue that results in scarring, characteristic of fibrotic liver disease. Liver fibrosis progresses from fatty liver disease, not all fatty liver disease patients develop fibrotic liver disease.

The Fibroscan device has an optional software module that attempts to quantify the attenuation of the shear wave as it travels away from the plane of deformation. Fibroscan refers to this measurement as CAP (Calculated Attenuation Parameter). The attenuation of the shear wave is thought to be related to the degree of liver steatosis (fat content). To date, the technique has demonstrated poor sensitivity, and is poorly correlated with quantitative MRI measures of liver fat. Furthermore, CAP measurements in obese patients are difficult to obtain and unreliable . Endra's technology aims to provide much more sensitive measurements of liver fat content at the point of care. The Endra device has the potential to quantify fat content as low as 5% (by volume). The system is interoperable with ultrasound and leverages B-mode ultrasound imaging to guide measurement location. Compared to Fibroscan's CAP, Endra's fatty liver measures are expected to be much more sensitive and reproducible based on anatomical guidance by ultrasound imaging.

ELIGIBILITY:
Inclusion Criteria:

* - Healthy volunteers which represent a range of genders, age, BMI and lifestyle.
* Must be over the age of 18.
* Must be proficient in English (reading/writing).

Exclusion Criteria:

* - Any metal or electronic implants including but not limited to pacemakers, metal clips, hips.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This feasibility study will recruit 25 healthy volunteers to undergo an ultrasound and thermoacoustic, and MRI examination of their liver while breathing normally, and during short breath-hold periods
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2023-08-08 (Actual); Study Completion 2023-08-08 (Actual)

PRIMARY OUTCOMES:
Fat concentration estimate | September 2019
  The purpose of the device is to measure the fat content of liver tissue to assist in the diagnosis of fatty liver disease.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Fenster, PhD, Principal Investigator — The University of Western Ontario
Locations (1):
- Aaron Fenster, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided